CLINICAL TRIAL: NCT02746237
Title: A Randomized, Double-blind, Placebo-controlled, Phase 1, First-in-human, Single-center, Safety, Tolerability, Ventricular Repolarization and Pharmacokinetic Study of Single and Multiple Ascending Doses of KAR5585 in Healthy Subjects
Brief Title: Single and Multiple Ascending Doses Clinical Pharmacology Study With KAR5585
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Karos Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: KAR5585-101
Record Dates: First submitted 2016-03-18; First posted 2016-04-21 (Estimated); Last update posted 2016-08-30 (Estimated); Status verified 2016-08

CONDITIONS: Pulmonary Arterial Hypertension
Keywords: Serotonin; Pulmonary Arterial Hypertension; Pharmacokinetics; Phase 1; Healthy Volunteers
MeSH Terms: conditions — Pulmonary Arterial Hypertension | interventions — rodatristat

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- KAR5585 (Experimental): KAR5585 Capsules
  Interventions: Drug: KAR5585 Capsules
- Placebo (Placebo Comparator): Placebo capsules
  Interventions: Drug: Placebo Capsules

INTERVENTIONS:
Drug: KAR5585 Capsules — Single and multiple ascending doses of KAR5585 (100 mg initial dose)
  Other Names: KAR5585
  Arms: KAR5585
Drug: Placebo Capsules — Single and multiple ascending doses of placebo (100 mg initial dose)
  Arms: Placebo

SUMMARY:
Safety, tolerability, pharmacokinetics (PK), cardiac conduction and food effect study on single and multiple ascending doses of KAR5585 in healthy adults.

DETAILED DESCRIPTION:
The purpose of this study is to explore the safety, tolerability, pharmacokinetics (PK), and cardiac conduction effects of single and multiple ascending doses of KAR5585 in healthy adults. Food effect will also be evaluated after a single-dose administration.

ELIGIBILITY:
Inclusion Criteria:

* Subject is able to read, write, and comprehend English at a sufficient level to understand study-related materials
* Subject is able to provide written informed consent and to comply with all study requirements and restrictions
* Subject is male or female and aged 18 to 65 years, inclusive, at the time of informed consent
* Subject is in good health as determined by the PI based on detailed medical history, physical examination, vital signs, clinical laboratory tests, ECGs, and other pre-dose evaluations
* Subject agrees to use a medically acceptable form of birth control from CRU admission until at least 30 days (female subject) or 90 days (male subject) after the last dose of study drug. Males will also not donate sperm from CRU admission until at least 90 days after the last dose of study drug. If a subject is not sexually active but becomes active during study participation, the subject agrees they and their partner will use a medically accepted form of contraception for the time specified. Medically acceptable forms of contraception are:

  * FDA-approved female hormonal contraceptives used consistently for 2 or more cycles before Screening, including oral contraceptives, intrauterine device (IUD), medroxyprogesterone acetate injection (Depo Provera®), hormonal implant (Norplant®, Implanon®, Nexplanon®), and vaginal ring (NuvaRing®)
  * Male condom plus spermicide
  * Male condom plus contraceptive sponge, foam, or jelly
  * Female condom plus spermicide
  * Diaphragm with spermicide plus male condom
  * Cervical cap with spermicide plus male condom
  * Surgical sterilization of the subject or partner (vasectomy for males, hysterectomy or bilateral oophorectomy for females)
  * Abstinence
* If female, subject agrees that a serum pregnancy test ([β hCG] beta human chorionic gonadotropin ) will be performed at Screening, on Day 2 (CRU admission), and at the last study visit and negative test results at Screening and CRU admission are required to be considered for study participation
* Subject has a body mass index (BMI) of 20 to 35 kg/m2, inclusive, and body weight < 120 kg at Screening

Exclusion Criteria:

* Subject currently uses tobacco or nicotine-containing products or has used such products within 6 months before CRU admission
* Subject has history or current evidence of any clinically significant cardiac, endocrinologic, hematologic, hepatobiliary, immunologic, metabolic, urologic, pulmonary, neurologic, dermatologic, psychiatric, renal, or other major disease, as determined by the PI
* Subject has a history of cancer within 5 years before CRU admission (excluding non-melanoma skin cancer)
* Subject has a history of autonomic dysfunction (eg, history of repeated dizziness, fainting, or symptomatic orthostatic hypotension)
* Subject has a history of risk factors for torsades de pointes, including unexplained syncope, known long QT syndrome, heart failure, myocardial infarction, angina, OR clinically significant abnormal laboratory assessments including hypokalemia, hypomagnesemia, or hypercalcemia OR has a family history of long QT syndrome or Brugada syndrome
* Subject has 1 or more clinically significant abnormal laboratory test values (as determined by the PI)
* Subject has an uninterpretable or abnormal screening ECG indicating a second- or third-degree atrioventricular block, or 1 or more of the following: QRS interval (ventricular depolarization) > 110 msec; a PR interval (atrioventricular conduction) > 220 msec, or QTc (corrected QT interval) of ≥ 450 msec (for male) or ≥ 470 msec (for female) or any rhythm other than sinus rhythm that is interpreted by the PI or a qualified designee to be clinically significant
* Subject has a resting heart rate (HR) of < 40 beats/min or > 90 beats/min at Screening or on CRU admission
* Subject has a sustained supine systolic blood pressure (BP) > 155 or < 90 mm Hg or a supine diastolic BP > 95 or < 50 mm Hg at Screening or upon CRU admission. Blood pressure in the supine position may be retested once and 'sustained' is defined as the parameter (either systolic or diastolic BP) being outside the stated limits at both assessments.
* Subject participates in another clinical trial or treatment with an investigational agent within 30 days or 5 half-lives, whichever is longer, before CRU admission
* Subject has a history of alcohol or drug abuse or dependence within 12 months before CRU admission, as determined by the PI
* Subject has a clinically significant infection within 3 months before CRU admission, as determined by the PI
* Subject has any condition that, in the opinion of the PI, would make the subject unsuitable for enrollment or could interfere with the subject's participation in or completion of the study
* Subject has a positive urine screen for prohibited drugs (cocaine, cannabinoids, nicotine [urine cotinine is the detection mechanism for nicotine], opiates, barbiturates, amphetamines, and benzodiazepines) or positive urine test for alcohol
* Subject has a positive blood screen for human immunodeficiency virus, hepatitis B surface antigen, or hepatitis C virus antibody at the Screening Visit
* Subject has had a known or suspected hypersensitivity or idiosyncratic reaction to the cellulose used in the placebo to be used in this study
* Subject has donated blood or any blood products within 3 months before Screening or plans to donate blood during or within 3 months after study completion
* Subject consumes an excessive amount of caffeine daily, defined as > 4 cups of coffee or equivalent per day. Subjects will abstain from caffeine consumption for 48 hours before dosing and while confined to the CRU.
* Subject has consumed or will consume any concomitant therapy; prescription or over-the-counter (OTC) medication; or nutritional, herbal, or vitamin supplements other than contraceptives (eg, oral, systemic) and ibuprofen (only if needed, maximum 2.4 g/day) from 14 days or 5 half-lives (whichever is longer) before dosing and while confined to the CRU
* For Part 2 only: Subject has consumed any food, juice, beverage, or medication (prescription or non-prescription) containing acetaminophen, alcohol, avocado, banana, caffeine, eggplant, kiwi fruit, nut (hickory nut, pecan, walnut), pineapple, plum, or tomato products within 48 hours before CRU admission

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 120 (Actual)
Dates: Start 2015-11; Primary Completion 2016-05 (Actual); Study Completion 2016-08 (Actual)

PRIMARY OUTCOMES:
Number of participants with abnormal physical exam results | From baseline to 4 days post-dose for single dose and baseline to 6 days post-dose for multiple doses
  Healthy adult volunteers receiving single and multiple doses of KAR5585 administered orally will be monitored for adverse events via physical examination.
Number of participants with abnormal hematology values | From baseline to 4 days post-dose for single dose and baseline to 6 days post-dose for multiple doses
  Healthy adult volunteers receiving single and multiple doses of KAR5585 administered orally will be monitored for adverse events via lab evaluation of hematology.
Number of participants with abnormal electrocardiogram results | From baseline to 4 days post-dose for single dose and baseline to 6 days post-dose for multiple doses
  Healthy adult volunteers receiving single and multiple doses of KAR5585 administered orally will be monitored for abnormal ECG results.
Number of participants with abnormal clinical chemistry values | From baseline to 4 days post-dose for single dose and baseline to 6 days post-dose for multiple doses
  Healthy adult volunteers receiving single and multiple doses of KAR5585 administered orally will be monitored for adverse events via lab evaluation of clinical chemistries.
Number of participants with abnormal urinalysis values | From baseline to 4 days post-dose for single dose and baseline to 6 days post-dose for multiple doses
  Healthy adult volunteers receiving single and multiple doses of KAR5585 administered orally will be monitored for adverse events via lab evaluation of urinalysis.

SECONDARY OUTCOMES:
Plasma area under the curve (AUC0-24) of prodrug KAR5585 and active inhibitor KAR5417 from time zero to 24 hours after dosing | From 0-24 hours on Days 1, 7 and 14
  Assessment of AUC 0-24 hours measured on Day 1, 7 and 14 when drug is dosed without a meal
Time to reach maximum observed plasma concentration (Tmax) of prodrug KAR5585 and active inhibitor KAR5417 | From 0-24 hours on Days 1, 7 and 14
  Assessment of Tmax measured on Day 1, 7 and 14 when drug is dosed without a meal
Plasma terminal elimination half- life (T1/2) of prodrug KAR5585 and active inhibitor KAR5417 | From 0-24 hours on Days 1, 7 and 14
  Assessment of T1/2 measured on Day 1, 7 and 14 when drug is dosed without a meal
Apparent volume of distribution (Vz/F) of prodrug KAR5585 and active inhibitor KAR5417 | From 0-24 hours on Days 1, 7 and 14
  Assessment of Vz/F measured on Day 1, 7 and 14 when drug is dosed without a meal
Maximum peak concentration (Cmax) of prodrug KAR5585 and active inhibitor KAR5417 | From 0-24 hours on Days 1, 7 and 14
  Assessment of Cmax measured on Day 1, 7 and 14 when drug is dosed without a meal
Serum levels of serotonin (ng/mL) | Days 1, 7 and 14
  Serum serotonin (5-HT) levels will be measured to evaluate the pharmacodynamic effects of KAR5585 administration
Urinary levels of 5-hydroxyindoleacetic acid(mg/24 hrs) | From 0-24 hours on Days 1, 7 and 14
  24 hour urine collection with analysis for 5-HIAA (5-hydroxyindoleacetic acid) levels.
Urinary levels of creatinine (gm/24 hrs) | From 0-24 hours on Days 1, 7 and 14
  24 hour urine collection with analysis for creatinine levels.
Urinary levels of 5-hydroxyindoleacetic acid normalized to creatinine (mg/gm) | From 0-24 hours on Days 1, 7 and 14
  24 hour urine collection with analysis for 5-HIAA (5-hydroxyindoleacetic acid). Urinary creatinine will be used to normalize urinary 5-HIAA levels: urinary 5-HIAA mg/gm creatinine
Plasma levels of 5-hydroxyindoleacetic acid (ng/mL) | Days 1, 7 and 14
  Plasma 5-HIAA (5-hydroxyindoleacetic acid) levels will be measured to evaluate the pharmacodynamic effects of KAR5585 administration
Plasma area under the curve (AUC0-24) of prodrug KAR5585 and active inhibitor KAR5417 from time zero to 24 hours after dosing | From 0-24hrs on Days 1, 7 and 14
  To determine the effect of food intake on the pharmacokinetics of KAR5585 and its active metabolite KAR5417, a cohort of patients will be studied after a single dose given fasting, followed by the same dose given with a high fat content food.
Time to reach maximum observed plasma concentration (Tmax) of prodrug KAR5585 and active inhibitor KAR5417 | From 0-24hrs on Days 1, 7 and 14
  To determine the effect of food intake on the pharmacokinetics of KAR5585 and its active metabolite KAR5417, a cohort of patients will be studied after a single dose given fasting, followed by the same dose given with a high fat content food.
Plasma terminal elimination half-life (T1/2) of prodrug KAR5585 and active inhibitor KAR5417 | From 0-24hrs on Days 1, 7 and 14
  To determine the effect of food intake on the pharmacokinetics of KAR5585 and its active metabolite KAR5417, a cohort of patients will be studied after a single dose given fasting, followed by the same dose given with a high fat content food.
Apparent volume of distribution (Vz/F) of prodrug KAR5585 and active inhibitor KAR5417 | From 0-24hrs on Days 1, 7 and 14
  To determine the effect of food intake on the pharmacokinetics of KAR5585 and its active metabolite KAR5417, a cohort of patients will be studied after a single dose given fasting, followed by the same dose given with a high fat content food.
Maximum peak concentration (Cmax) of prodrug KAR5585 and active inhibitor KAR5417 | From 0-24hrs on Days 1, 7 and 14
  To determine the effect of food intake on the pharmacokinetics of KAR5585 and its active metabolite KAR5417, a cohort of patients will be studied after a single dose given fasting, followed by the same dose given with a high fat content food.

CONTACTS AND LOCATIONS:
Overall Officials: Carlos Sanabria, MD, Principal Investigator — Spaulding Clinical
Locations (1):
- Spaulding Clinical, West Bend, Wisconsin, United States

IPD SHARING:
Plan to Share IPD: No